CLINICAL TRIAL: NCT06773780
Title: Transcatheter Aortic Valve Implantation: Comparison of the Effects of Ultrasound-Guided Pericapsular Nerve Group Block and Fascia Iliaca Block on Postoperative Analgesia Management - A Randomized, Prospective Study
Brief Title: Transcatheter Aortic Valve Implantation: Comparison of the Effects of Ultrasound-Guided Pericapsular Nerve Group Block and Fascia Iliaca Block on Postoperative Analgesia Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TAVİ PENG VS FİB
Record Dates: First submitted 2024-12-27; First posted 2025-01-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Pericapsular Nerve Group Block; Fascia Iliaca Block
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local infiltration (Active Comparator): Under sterile conditions, 30 ml of 0.25% bupivacaine will be applied to the targeted infiltration area.
  Interventions: Drug: local infiltration
- PENG (Active Comparator): For the PENG block, the patient is placed in the supine position, and a sterile-covered convex ultrasound probe is positioned transversely over the anterior inferior iliac spine. After identifying the femoral artery, iliopubic eminence, and psoas muscle, the needle is advanced in-plane between the pubic ramus and psoas tendon, and 30 mL of 0.25% bupivacaine is injected.
  Interventions: Drug: PENG
- FİB (Active Comparator): For the FIB, with the patient's legs slightly externally rotated, a high-frequency ultrasound probe is placed along the inguinal ligament. The needle is advanced beneath the fascia iliaca, and 30 mL of 0.25% bupivacaine is injected under ultrasound guidance.
  Interventions: Drug: FİB

INTERVENTIONS:
Drug: local infiltration — The block procedure will be performed before the surgical procedure, following the induction of sedoanalgesia. Under sterile conditions, 30 mL of 0.25% bupivacaine will be administered to the targeted infiltration area. The local anesthetic will be specifically applied around the arterial and venous puncture sites.
  Arms: Local infiltration
Drug: PENG — With the patient in the supine position, a convex ultrasound (US) probe (4-8 MHz, Vivid Q) will be covered with a sterile sheath. An 80-mm block needle (Braun 360°) will be used. The probe will be placed transversely over the anterior inferior iliac spine. Subsequently, the probe will be rotated 45 degrees to visualize the pubic ramus. Once the femoral artery, iliopubic eminence, and psoas muscle are identified under ultrasound guidance, the needle will be advanced using an in-plane technique and positioned between the pubic ramus and the psoas tendon. After confirming the block site with 5 mL of saline, 30 mL of 0.25% bupivacaine will be injected as the local anesthetic.
  Arms: PENG
Drug: FİB — The patient's legs will be positioned slightly externally rotated. A high-frequency ultrasound probe will be placed transversely along the inguinal ligament. Under ultrasound guidance, the femoral artery, iliopsoas muscle, and fascia iliaca will be identified. The needle will be advanced parallel to the ultrasound probe using the in-plane technique and positioned beneath the fascia iliaca. After confirming negative aspiration, 30 mL of 0.25% bupivacaine will be injected, and the spread of the solution beneath the fascia iliaca will be verified using ultrasound.
  Arms: FİB

SUMMARY:
Aortic Stenosis (AS) is the most common valvular pathology, particularly prevalent in advanced age, and Transcatheter Aortic Valve Implantation (TAVI) has become a crucial treatment option for high-risk patients who are not suitable for surgery. This minimally invasive approach has demonstrated successful clinical outcomes in patients deemed ineligible for surgical procedures.

Patient selection criteria and advancements in operative techniques are critical for achieving successful TAVI outcomes. While the transfemoral approach is the most commonly used method, alternative techniques such as transapical, transaxillary, transcarotid, and transaortic approaches are also available.

The Pericapsular Nerve Group Block (PENG) targets the femoral and accessory obturator nerves, providing analgesia to the anterior hip without causing motor block. The Fascia Iliaca Block (FIB), on the other hand, provides broader analgesic coverage by affecting the lateral femoral cutaneous, obturator, and femoral nerves.

This study aims to compare PENG block, FIB, and local infiltration anesthesia in TAVI patients regarding sedation requirements during the procedure and postoperative analgesia management. Additionally, pain scores, motor block presence, opioid consumption, and side effects will be assessed. The study seeks to identify optimal strategies to enhance patient comfort and safety during TAVI procedures.

DETAILED DESCRIPTION:
Aortic Stenosis (AS) is the most common valvular pathology, affecting 2% to 4% of individuals over the age of 75. Surgical Aortic Valve Replacement (SAVR) has long been considered the first-line recommendation for AS treatment. However, due to advanced age and the increasing prevalence of severe comorbidities, more than one-third of high-risk and severely symptomatic AS patients are deemed physiologically unsuitable for major surgical interventions.

This situation has led to the development and implementation of Transcatheter Aortic Valve Implantation (TAVI) as an alternative intervention for high-risk patients and those deemed unsuitable for surgery. This shift towards minimally invasive procedures has resulted in revolutionary improvements in clinical outcomes, particularly for AS patients previously considered ineligible for surgery.

Advances in patient selection criteria and operative techniques have made significant contributions to the success of TAVI. Both retrograde and anterograde operative approaches can be employed during the TAVI procedure. While the transfemoral approach remains the most commonly used technique, alternative methods such as transapical, transaxillary, transcarotid, and transaortic approaches are also available. The choice of operative technique largely depends on patient-specific anatomical features and existing comorbidities.

Pericapsular Nerve Group Block (PENG Block) The increasing use of ultrasound (US) in anesthetic practice has facilitated the frequent application of US-guided nerve blocks. The Pericapsular Nerve Group Block (PENG Block) is a novel fascial block first described by Arango et al. In this technique, local anesthetic is injected between the pubic ramus and the psoas tendon, targeting the femoral and accessory obturator nerves to provide effective analgesia for the anterior hip region.

The PENG block has the advantage of not causing motor block. Its superficial applicability makes it a safe and effective method. Radiological and cadaver studies have shown that high-volume local anesthetic injections can also block the lateral femoral cutaneous, genitofemoral, obturator, and femoral nerves, enabling total hip analgesia.

Fascia Iliaca Block (FIB) The Fascia Iliaca Block (FIB) is an effective fascial block technique capable of simultaneously affecting multiple nerves. This block aims to anesthetize the lateral femoral cutaneous, obturator, and femoral nerves, providing broad analgesic coverage. FIB is performed away from critical inguinal neurovascular structures, enhancing its reliability. It is particularly preferred in pain management scenarios, such as acute hip fractures, and is considered a safe option for these clinical situations.

Aim of the Study This prospective, randomized study aims to compare the sedation requirements during the procedure and the postoperative analgesia management in TAVI patients undergoing PENG block, FIB, or local infiltration anesthesia. The primary objective is to evaluate the sedation needs of patients during the procedure. The secondary objectives include comparing postoperative pain scores (Numerical Rating Scale - NRS), the presence of quadriceps motor block (paretic or paralytic knee extension), opioid consumption, and opioid-related side effects (e.g., allergic reactions, nausea, vomiting).

This study aims to analyze the efficacy and safety of different analgesia methods, contributing to the identification of optimal strategies to enhance patient comfort and safety during TAVI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for TAVİ
* aged between 18 and 85 years,
* American Society of Anesthesiology (ASA) physical status II-IV

Exclusion Criteria:

* History of bleeding diathesis.
* Use of anticoagulant therapy.
* History of chronic pain prior to surgery.
* Multiple trauma.
* Conditions where pain assessment cannot be performed (e.g., dementia).
* Patients operated under spinal or epidural anesthesia.
* Presence of infection in the region where the block will be applied.
* Refusal to consent to the procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of sedation requirements and the amount of sedative medication used during the TAVI procedure will be evaluated. | during the procedure
  The amounts of anesthetic and opioid drugs used during the procedure will be compared.

SECONDARY OUTCOMES:
the aim of this study is to compare postoperative NRS (Numerical Rating Scale) pain scores of the patients between the groups. | first 24 hours after the operation
  The NRS is an 11-point scale. Zero means 'no pain', 10 means 'the most severe pain imaginable'. NRS scores at rest and during mobilization are evaluated and recorded in the postoperative recovery unit at 3, 6, 12, 18 and 24 hours. If the NRS score is ≥ 4, 1 mg kg-1 IV tramadol is administered as a rescue analgesic.
The aim of this study is to compare opioid-related side effects (such as nausea, vomiting, respiratory depression) of the patients between the groups. | first 24 hours after the operation
  It will be evaluated whether there are any opioid-related side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544